CLINICAL TRIAL: NCT02101112
Title: Relative Bioavailability of Crushed Apixaban Tablets Administered With Water or Apple Sauce Compared With Intact Tablet in Healthy Subjects
Brief Title: Bioavailability of Apixaban Crushed Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV185-292
Record Dates: First submitted 2014-03-28; First posted 2014-04-01 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apixaban, 10 mg (whole tablets) (Experimental): Participants received a single dose of apixaban, 10 mg, given orally as 2 5-mg whole commercial tablets (reference)
  Interventions: Drug: Apixaban
- Apixaban, 10 mg (crushed and suspended in water) (Experimental): Participants received a single dose of apixaban, 10 mg, given by mouth as 2 5-mg whole commercial tablets crushed and suspended in 30 mL of water
  Interventions: Drug: Apixaban
- Apixaban, 10 mg (crushed and mixed with applesauce) (Experimental): Participants received a single dose of 10 mg, given by mouth as 2 5-mg apixaban commercial tablets crushed and mixed with 30 g of applesauce
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis®

SUMMARY:
The purpose of this study is to determine whether the bioavailability of apixaban crushed tablets suspended in water or mixed with applesauce is similar to the bioavailability of apixaban whole tablets administered orally.

DETAILED DESCRIPTION:
This study will investigate the bioavailability of apixaban administered as crushed tablets suspended in water and as crushed tablets mixed with applesauce compared with that of whole tablets. The study results may allow enhancement of the apixaban label to include alternative methods of apixaban administration, which may be of benefit to patients who have difficulty swallowing.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal in findings of medical history, physical examination, electrocardiograms, vital signs, and clinical laboratory tests.
* Women of childbearing potential allowed. Must be following highly effective methods of contraception

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of significant head injury within the last 2 years, including individuals with base of skull fractures
* Any major surgery within 4 weeks of study drug administration or anticipated within 2 weeks after completion of the study
* Any gastrointestinal (GI) surgery or GI disease that could impact absorption of study drug
* History of Gilbert's Syndrome
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access
* Use of tobacco- or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to study drug administration
* Any laboratory test results outside of the range of normal, confirmed by repeat results of:

  * Platelet count <150,000 cells/µL
  * Activated partial thromboplastin time >upper limit of normal (ULN)
  * International normalized ratio >ULN
  * Alanine aminotransferase >ULN
  * Aspartate aminotransferase >ULN
  * Total bilirubin >ULN
  * Serum creatinine ≥1.5 mg/dL
  * Hemoglobin <lower limit of normal (LLN)
  * Hematocrit <LLN

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Song Y, Chang M, Suzuki A, Frost RJ, Kelly A, LaCreta F, Frost C. Evaluation of Crushed Tablet for Oral Administration and the Effect of Food on Apixaban Pharmacokinetics in Healthy Adults. Clin Ther. 2016 Jul;38(7):1674-1685.e1. doi: 10.1016/j.clinthera.2016.05.004. Epub 2016 Jun 10. PMID 27292282
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 69 participants enrolled, 33 participants randomized. 36 participants were enrolled but not randomized. Reasons for non-randomization include 30 participants no longer met study criteria, 4 participants withdrew consent, 2 participants were not needed for the study.
Groups:
- Treatment A Then Treatment B Then Treatment C; Treatment A Then Treatment C Then Treatment B; Treatment B Then Treatment C Then Treatment A; Treatment B Then Treatment A Then Treatment C; Treatment C Then Treatment A Then Treatment B; Treatment C Then Treatment B Then Treatment A: Treatment A = Apixaban, 10 mg (Whole Tablets); Participants received a single dose of apixaban, 10 mg, given orally as two 5-mg whole commercial tablets.
  Treatment B = Apixaban, 10 mg (Crushed and Suspended in Water); Participants received a single dose of apixaban, 10 mg, given by mouth as two 5-mg whole commercial tablets crushed and suspended in 30 mL of water.
  Treatment C = Apixaban, 10 mg (Crushed and Mixed With Applesauce); Participants received a single dose of 10 mg, given by mouth as two 5-mg apixaban commercial tablets crushed and mixed with 30 g of applesauce
  This was a 3-period, 3-treatment crossover study. Each participant received (orally) a single-dose of apixaban 10 mg (two 5-mg tablets) crushed and suspended in 30 mL water and a single-dose of apixaban 10 mg (two 5-mg tablets) crushed and mixed with 30 g applesauce according to a randomization schedule. Each participant underwent a washout of at least 4 days before receiving the next scheduled treatment.
Period: Overall Study
Arm/Group | Treatment A Then Treatment B Then Treatment C | Treatment A Then Treatment C Then Treatment B | Treatment B Then Treatment C Then Treatment A | Treatment B Then Treatment A Then Treatment C | Treatment C Then Treatment A Then Treatment B | Treatment C Then Treatment B Then Treatment A
Started | 6 | 5 | 6 | 5 | 6 | 5
Completed | 6 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Apixaban, 10 mg (Whole Tablets): This was a 3-period, 3-treatment crossover study. Each participant received (orally) a single-dose of apixaban 10 mg (two 5-mg tablets) crushed and suspended in 30 mL water and a single-dose of apixaban 10 mg (two 5-mg tablets) crushed and mixed with 30 g applesauce according to a randomization schedule. Each participant underwent a washout of at least 4 days before receiving the next scheduled treatment.
Arm/Group | Apixaban, 10 mg (Whole Tablets)
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Weight [Mean (Standard Deviation); unit: kilograms] | 77.40 (7.933)
Height [Mean (Standard Deviation); unit: centimeters] | 172.13 (8.322)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter^2] | 26.14 (2.166)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Apixaban
Description: Maximum observed plasma concentration (Cmax) measured in nanograms per milliliter (ng/mL)
Time Frame: Days 1, 5, and 9 predose and 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60 and 72 hours post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Apixaban, 10 mg (Whole Tablets): Participants received a single dose of apixaban, 10 mg, given orally as two 5-mg whole commercial tablets.
- Apixaban, 10 mg (Crushed and Suspended in Water): Participants received a single dose of apixaban, 10 mg, given by mouth as two 5-mg whole commercial tablets crushed and suspended in 30 mL of water.
- Apixaban, 10 mg (Crushed and Mixed With Applesauce): Participants received a single dose of 10 mg, given by mouth as two 5-mg apixaban commercial tablets crushed and mixed with 30 g of applesauce
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
ng/mL | 236 [217 to 256] | 249 [232 to 266] | 186 [174 to 199]
Statistical Analysis 1: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Suspended in Water); Apixaban, 10 mg (crushed and suspended in water) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 1.054, 90% CI 2-sided [0.994 to 1.118]
Statistical Analysis 2: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Mixed With Applesauce); Apixaban, 10 mg (crushed and mixed with applesauce) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.788, 90% CI 2-sided [0.741 to 0.839]

2. Primary Outcome: Adjusted Geometric Mean of Area Under the Plasma Concentration-time Curve (AUC) From Time Zero Extrapolated to Infinite Time [AUC(INF)] of Apixaban
Description: Area Under the Plasma Concentration-time Curve (AUC) From Time of Zero Extrapolated to Infinite Time (INF) [AUC (INF)] is measured as nanograms multiplied by hours per milliliter (ng*h/mL)
Time Frame: Days 1, 5, and 9 predose and 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, and 72 hours post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
ng*h/mL | 2461 [2273 to 2664] | 2528 [2375 to 2692] | 2055 [1915 to 2206]
Statistical Analysis 1: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Suspended in Water); Apixaban, 10 mg (crushed and suspended in water) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 1.027, 90% CI 2-sided [0.981 to 1.076]
Statistical Analysis 2: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Mixed With Applesauce); Apixaban, 10 mg (crushed and mixed with applesauce) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.835, 90% CI 2-sided [0.797 to 0.875]

3. Primary Outcome: Adjusted Geometric Mean of Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Apixaban
Description: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Quantifiable Concentration [AUC (0-T)] is measured as nanograms multiplied by hours per milliliter (ng*h/mL)
Time Frame: Days 1, 5, and 9 predose and 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, and 72 hours post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
ng*h/mL | 2423 [2238 to 2623] | 2488 [2336 to 2651] | 2015 [1876 to 2165]
Statistical Analysis 1: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Suspended in Water); Apixaban, 10 mg (crushed and suspended in water) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 1.027, 90% CI 2-sided [0.981 to 1.075]
Statistical Analysis 2: Comparison: Apixaban, 10 mg (Whole Tablets) vs Apixaban, 10 mg (Crushed and Mixed With Applesauce); Apixaban, 10 mg (crushed and mixed with applesauce) vs. Apixaban, 10 mg (whole tablets); Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.832, 90% CI 2-sided [0.794 to 0.871]

4. Secondary Outcome: Number of Participants With Serious Adverse Events, Death, or Discontinuation Due to Adverse Events by Study Completion
Description: Adverse Event (AE) = any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious Adverse Event (SAE)= a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Randomization to May 2014; approximately 6 weeks
Population: All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
participants
  Deaths | 0 | 0 | 0
  SAEs | 0 | 0 | 0
  Drug-related AEs | 0 | 1 | 0
  Discontinuation due to AE | 0 | 1 | 0

5. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Apixaban
Description: Time of maximum observed plasma concentration (Tmax) measured in hours (h)
Time Frame: Days 1, 5 and 9 pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12 24, 36, 48, 60 and 72 hrs post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Median (Full Range); unit: hours
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
hours | 2.00 [1.00 to 5.00] | 2.00 [0.583 to 4.00] | 2.00 [1.00 to 4.00]

6. Secondary Outcome: Terminal Plasma Half-life (T-HALF) of Apixaban
Description: Terminal plasma half-life (T-HALF) was derived from plasma concentration versus time data. T-HALF was the time required for one half of the total amount of administered drug to be eliminated from the body.
Time Frame: Days 1, 5 and 9 pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12 24, 36, 48, 60 and 72 hrs post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 33 | 32
hours | 12.4 (5.39) | 12.2 (5.19) | 12.5 (5.05)

7. Secondary Outcome: Relative Bioavailability (Frel) of Apixaban
Description: Frel is calculated using the treatment ratio of AUC(INF) where the denominator is the AUC(INF) of the reference therapy, 10mg of Apixaban (whole tablet).
Time Frame: Days 1, 5 and 9 pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12 24, 36, 48, 60 and 72 hrs post dose
Population: All evaluable pharmacokinetic (PK) participants who were treated with apixaban
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Number analyzed (Participants) | 32 | 32
ratio | 1.03 (24) | 0.836 (20)

ADVERSE EVENTS:
Time Frame: Day 1 to May 2014; approximately 6 weeks F
Description: Study initiated: March 2014; Study Completion: May 2014
Arm/Group | Apixaban, 10 mg (Whole Tablets) | Apixaban, 10 mg (Crushed and Suspended in Water) | Apixaban, 10 mg (Crushed and Mixed With Applesauce)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.